CLINICAL TRIAL: NCT04297852
Title: The Function of Nutrition Rich Vegan Drink on Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Per Bendix Jeppesen (Other)
Collaborators: Future Food Innovation (Industry)
Responsible Party: Sponsor-Investigator, Per Bendix Jeppesen, Associate. Prof, PhD., University of Aarhus
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: VEGJUICE
Record Dates: First submitted 2019-02-21; First posted 2020-03-06 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Recovery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vegan drink (Active Comparator): Treatment group
  Interventions: Dietary Supplement: Vegan drink
- Control (Placebo Comparator): Placebo group
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Vegan drink — Vegan based drink containing vegetables, fruits and plant oils. Dose: 500 mL a day
  Arms: Vegan drink
Dietary Supplement: Control — Placebo drink Dose: 500 mL a day
  Arms: Control

SUMMARY:
The aim of this project, would be to develop a new formula, with high nutrition content on a vegan basis. The investigators expect to produce this novel vegan-based juice product, which does not exist on the marked today. The juice would consist of different selected varieties of vegetables and fruits. Beside the vegetables, the juice will also contain plant oils to increase the calorie level, as well as a protein sources containing amino acids with high anabolic effects.

The products will be tested in an intervention study on patients with inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 85 years old
* Diagnosed with or show signs of UC or Crohns disease
* Mild symptoms i.e intestinal symptoms
* Has had the same medicin the previous week before starting in the study

Exclusion Criteria:

* Food or vegetable allergi
* Cognitive diseases e.g alzheimers or dementia
* Has diabetes requiring insulin or GLP-1 analog treatment (NB: No does include T2D patients, taking tablets or other diabetes therapy)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Inflammatory factors | 3 weeks
  F-calprotectin

CONTACTS AND LOCATIONS:
Overall Officials: Per B Jeppesen, Prof, Principal Investigator — Department of clinical medicin
Locations (1):
- Aarhus university, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No